CLINICAL TRIAL: NCT02707601
Title: A Phase 3b Randomized, Open-label, Controlled Study of the Efficacy, Safety and Tolerability of 12 Weeks of Ledipasvir/Sofosbuvir (LDV/SOF) Treatment for HIV/HCV Co-infected Subjects Who Switch to Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) or Emtricitabine/Rilpivirine/Tenofovir Alafenamide (F/R/TAF) Prior to LDV/SOF HCV Treatment, the HIV/HCV Co-STARs Study (Co-infection Treatment With Single Tablet Antiviral Regimens)
Brief Title: Efficacy, Safety, and Tolerability of Ledipasvir/Sofosbuvir (LDV/SOF) Treatment for HIV/HCV Co-infected Participants Who Switch to Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) or Emtricitabine/Rilpivirine/Tenofovir Alafenamide (F/R/TAF) Prior to LDV/SOF HCV Treatment
Acronym: Co-STARs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-366-1992; 2014-004545-27 (EudraCT Number)
Record Dates: First submitted 2016-03-09; First posted 2016-03-14 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-09

CONDITIONS: HIV-1 Infection; HCV Infection
Keywords: HIV; HCV; Antiretroviral therapy; HCV direct acting antiviral(s) (DAA)
MeSH Terms: conditions — Hepatitis C | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- E/C/F/TAF + LDV/SOF (Experimental): Part 1: Participants will switch from 2 nucleoside reverse transcriptase inhibitors (NRTI) plus a third agent to E/C/F/TAF.
  Part 2: After 8 weeks of E/C/F/TAF treatment, the participants maintaining HIV-1 RNA < 50 copies/mL will start receiving LDV/SOF for 12 weeks and continue their HIV treatment until the end of the study.
  Interventions: Drug: E/C/F/TAF; Drug: LDV/SOF
- F/R/TAF + LDV/SOF (Experimental): Part 1: Participants will switch from 2 NRTI plus a third agent to F/R/TAF.
  Part 2: After 8 weeks of F/R/TAF treatment, the participants maintaining HIV-1 RNA < 50 copies/mL will start receiving LDV/SOF for 12 weeks and continue their HIV treatment until the end of the study.
  Interventions: Drug: F/R/TAF; Drug: LDV/SOF

INTERVENTIONS:
Drug: E/C/F/TAF — 150/150/200/10 mg fixed dose combination (FDC) tablet administered orally once daily
  Other Names: Genvoya®
  Arms: E/C/F/TAF + LDV/SOF
Drug: F/R/TAF — 200/25/25 mg FDC tablet administered orally once daily
  Other Names: Odefsey®
  Arms: F/R/TAF + LDV/SOF
Drug: LDV/SOF — 90/400 mg FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977

SUMMARY:
This study will evaluate efficacy of ledipasvir/sofosbuvir (LDV/SOF) and safety and tolerability of switching to elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) or emtricitabine/rilpivirine/tenofovir alafenamide (F/R/TAF) from the current antiretroviral (ARV) therapy and in virologically-suppressed, HIV-1/HCV co-infected participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic genotype (GT) 1, HCV infected, male and non-pregnant/ non-lactating female individuals, without cirrhosis, treatment-naive or treatment-experienced with interferon (IFN) +/- ribavirin (RBV) +/- HCV protease inhibitor (PI).
* Compensated cirrhotic individuals must be HCV treatment-naive.
* No prior treatments with NS5A and NS5B or any HCV direct acting antivirals, except boceprevir, telaprevir and simeprevir, in combination with IFN and RBV
* Currently on an ARV regimen (2 NRTI + a third agent) without change for 6 months prior to screening.
* Documented plasma HIV-1 RNA levels < 50 copies/mL (or undetectable HIV-1 RNA level according to the local assay being used if the limit of detection is ≥ 50 copies/mL) for ≥ 6 months preceding the screening visit. After reaching HIV-1 RNA < 50 copies/mL, single values ("blips") of HIV-1 RNA ≥ 50 copies/mL followed by resuppression is allowed.
* For individuals with 3 or more prior ARV regimens, a regimen history should be provided for approval by the Sponsor.

  * Note: Individuals that changed from TDF to TAF less than 6 months ago will be eligible as long as the TDF/ TAF change was the only change to the regimen.
* Plasma HIV-1 RNA level < 50 copies/mL at the screening visit
* Have no documented resistance to any of the HIV study agents at time in the past, including but not limited to the reverse transcriptase resistance mutations K65R, K70E, K101E/P, E138A/G/K/R/Q, V179L, Y181C/I/V, M184V/I, Y188L, H221Y, F227C, M230I/L, the combination of K103N+L100I, or 3 or more thymidine analog associated mutations (TAMs) that include M41L or L210W (TAMs are M41L, D67N, K70R, L210W, T215Y/F, K219Q/E/N/R). If a historical genotype prior to first ARV is not available or individual had 3 or more prior ARV regimens, individual will have proviral genotype analysis for archived resistance prior to Day 1.
* No history of HIV virologic failure
* No evidence of Hepatitis B infection
* Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min as estimated by Cockcroft-Gault formula

Note: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (43):
- United States (42):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Spectrum Medical Group, Phoenix, Arizona
  - Mills Clinical Research, Los Angeles, California
  - Peter J Ruane MD Inc, Los Angeles, California
  - University of California Davis, Sacramento, California
  - University of California San Diego, San Diego, California
  - Kaiser Permanente, San Francisco, California
  - The George Washington University Medical Center, Washington D.C., District of Columbia
  - Whitman-Walker Health, Washington D.C., District of Columbia
  - Community AIDS Network, Clearwater, Florida
  - Gary Richmond, MD, PA, Inc., Fort Lauderdale, Florida
  - Therafirst Medical Center, Fort Lauderdale, Florida
  - Midway Immunology & Research Center, LLC, Ft. Pierce, Florida
  - University of Miami, Miami, Florida
  - AIDS Healthcare Foundation, Miami, Florida
  - AIDS Healthcare Foundation, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - St. Josephs Comprehensive Research Institute, Tampa, Florida
  - Triple O Research Institute PA, West Palm Beach, Florida
  - Rowan Tree Medical PA, Wilton Manors, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Chatham County Health Department, Savannah, Georgia
  - The CORE Foundation, Chicago, Illinois
  - Be Well Medical Center, Berkley, Michigan
  - Kansas City Free Health Clinic, Kansas City, Missouri
  - Saint Michael's Medical Center, Newark, New Jersey
  - Weill Cornell Medical College, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Lehigh Valley Health Network, Network Office of Research and Innovation, Allentown, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Central Texas Clinical Research, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Gordon E. Crofoot MD PA, Houston, Texas
  - Therapeutics Concepts, PA, Houston, Texas
  - Clinical Alliance for Research & Education, Annandale, Virginia
  - Peter Shalit MD, Seattle, Washington
  - Southern Cal, Spokane, Washington
  - Community Health Care, Tacoma, Washington
- Clinical Research Puerto Rico Inc, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Ramgopal M, Jain M, Hinestrosa F, Asmuth D, Huhn G, Slim J, et al. HIV-1/HCV Coinfection Treatment with Single-Tablet Antiviral Regimens (CoSTARs): 12 Weeks of Ledipasvir/Sofosbuvir (LDV/SOF) after Randomized Switch to Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) or Rilpivirine/F/TAF (R/F/TAF) [Poster LB-12]. AASLD: The Liver Meeting 2017 20-24 October; Washington DC.
- [Result] Huhn G, Jain M, Hinestrosa F, Asmuth D, Huhn G, Slim J, et al. HIV-1/HCV Coinfection Treatment with Single-Tablet Antiviral Regimens (CoSTARs): 12 Weeks of Ledipasvir/Sofosbuvir (LDV/SOF) after Randomized Switch to Elvitegravir/Cobicistat/ Emtricitabine/Tenofovir Alafenamide (E/C/F/TAF) or Rilpivirine/F/TAF (R/F/TAF) [Poster PE16/52]. European AIDS Conference 2017 25-27 October; Milan Italy.
- [Derived] Huhn GD, Ramgopal M, Jain MK, Hinestrosa F, Asmuth DM, Slim J, Goldstein D, Applin S, Ryu JH, Jiang S, Cox S, Das M, Nguyen-Cleary T, Piontkowsky D, Guyer B, Rossaro L, Haubrich RH. HIV/HCV therapy with ledipasvir/sofosbuvir after randomized switch to emtricitabine-tenofovir alafenamide-based single-tablet regimens. PLoS One. 2020 Jan 29;15(1):e0224875. doi: 10.1371/journal.pone.0224875. eCollection 2020. PMID 31995556

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 01 April 2016. The last study visit occurred on 29 September 2017.
Pre-assignment Details: 259 participants were screened.
Groups:
- E/C/F/TAF + LDV/SOF: Part 1: Participants received elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) 150/150/200/10 mg orally once daily with food for 8 weeks. At Week 8, participants who tolerated the switch to E/C/F/TAF and maintained HIV-1 RNA < 50 copies/mL continued to Part 2 of the study.
  Part 2: Participants continued receiving E/C/F/TAF 150/150/200/10 mg orally once daily with food until the end of the study and received ledipasvir/sofosbuvir (LDV/SOF) 90/400 mg orally once daily with or without food for 12 weeks (until Week 20).
- F/R/TAF + LDV/SOF: Part 1: Participants received emtricitabine/rilpivirine/tenofovir alafenamide (F/R/TAF) 200/25/25 mg orally once daily with food for 8 weeks. At Week 8, participants who tolerated the switch to F/R/TAF and maintained HIV-1 RNA < 50 copies/mL continued to Part 2 of the study.
  Part 2: Participants continued receiving F/R/TAF 200/25/25 mg orally once daily with food until the end of the study and received LDV/SOF 90/400 mg orally once daily with or without food for 12 weeks (until Week 20).
Period: Overall Study
Arm/Group | E/C/F/TAF + LDV/SOF | F/R/TAF + LDV/SOF
Started | 76 | 74
Completed | 72 | 70
Not Completed | 4 | 4
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Investigator's Discretion | 1 | 0
Not completed — Withdrew Consent | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Participants Randomized but Not Treated | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug (E/C/F/TAF, F/R/TAF, or LDV/SOF).
Groups:
- E/C/F/TAF + LDV/SOF: Part 1: Participants received E/C/F/TAF 150/150/200/10 mg orally once daily with food for 8 weeks. At Week 8, participants who tolerated the switch to E/C/F/TAF and maintained HIV-1 RNA < 50 copies/mL continued to Part 2 of the study.
  Part 2: Participants continued receiving E/C/F/TAF 150/150/200/10 mg orally once daily with food until the end of the study and received LDV/SOF 90/400 mg orally once daily with or without food for 12 weeks (until Week 20).
- F/R/TAF + LDV/SOF: Part 1: Participants received F/R/TAF 200/25/25 mg orally once daily with food for 8 weeks. At Week 8, participants who tolerated the switch to F/R/TAF and maintained HIV-1 RNA < 50 copies/mL continued to Part 2 of the study.
  Part 2: Participants continued receiving F/R/TAF 200/25/25 mg orally once daily with food until the end of the study and received LDV/SOF 90/400 mg orally once daily with or without food for 12 weeks (until Week 20).
- Total: Total of all reporting groups
Arm/Group | E/C/F/TAF + LDV/SOF | F/R/TAF + LDV/SOF | Total
Number analyzed (Participants) | 74 | 74 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (9.5) | 52 (9.9) | 51 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 22 | 38
  Male | 58 | 52 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 14 | 27
  Not Hispanic or Latino | 61 | 59 | 120
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black | 30 | 31 | 61
  White | 41 | 37 | 78
  Native Hawaiian or Pacific Islander | 0 | 2 | 2
  Other | 2 | 3 | 5
  American Indian or Alaska Native | 0 | 1 | 1
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 25 | 14 | 39
  ≥ 800,000 IU/mL | 49 | 60 | 109
HIV-1 RNA Category [Count of Participants; unit: Participants]
  < 50 copies/mL | 73 | 74 | 147
  ≥ 50 copies/mL | 1 | 0 | 1
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.0 (1.07) | 6.3 (0.74) | 6.2 (0.92)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HCV RNA < LLOQ at 12 Weeks After Discontinuation of LDV/SOF Treatment (SVR12)
Description: Sustained Virologic Response (SVR12) was defined as HCV RNA < the lower limit of quantitation (LLOQ) at 12 weeks after stopping LDV/SOF treatment.
Time Frame: HCV Posttreatment Week 12
Population: HCV Full Analysis Set: participants who were randomized into the study and received at least 1 dose of HCV study drug, LDV/SOF.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | E/C/F/TAF + LDV/SOF | F/R/TAF + LDV/SOF
Number analyzed (Participants) | 72 | 72
percentage of participants | 98.6 [92.5 to 100.0] | 95.8 [88.3 to 99.1]
Statistical Analysis 1: Comparison: E/C/F/TAF + LDV/SOF; Test type: Superiority; p = 0.002, Binomial test — The p-value is obtained from the 2-sided exact 1-sample binomial test for the superiority over the performance goal of 88%
Statistical Analysis 2: Comparison: F/R/TAF + LDV/SOF; Test type: Superiority; p = 0.042, Binomial test — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at 4 Weeks After Discontinuation of LDV/SOF Treatment (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping LDV/SOF treatment.
Time Frame: HCV Posttreatment Week 4
Population: HCV Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | E/C/F/TAF + LDV/SOF | F/R/TAF + LDV/SOF
Number analyzed (Participants) | 72 | 72
percentage of participants | 98.6 [92.5 to 100.0] | 98.6 [92.5 to 100.0]
Statistical Analysis 1: Comparison: E/C/F/TAF + LDV/SOF; Test type: Superiority; p = 0.002, Binomial test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: F/R/TAF + LDV/SOF; Test type: Superiority; p = 0.002, Binomial test — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL (Virologic Failure) 24 Weeks After Start of the F/TAF-Based Regimen Using Modified FDA Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA ≥ 50 copies/mL 24 weeks after start of the F/TAF-based regimen were analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: 24 weeks after start of HIV treatment
Population: HIV Full Analysis Set: participants who were randomized into the study and received at least 1 dose of HIV study drug, E/C/F/TAF or F/R/TAF.
Measure: Number; unit: percentage of participants
Arm/Group | E/C/F/TAF + LDV/SOF | F/R/TAF + LDV/SOF
Number analyzed (Participants) | 74 | 74
percentage of participants | 1.4 | 1.4
Statistical Analysis 1: Comparison: E/C/F/TAF + LDV/SOF vs F/R/TAF + LDV/SOF; Test type: Other; p = 1.00, Fisher exact test; Difference in Percentages = 0.0, 95% CI 2-sided [-6.1 to 6.1] — The differences in percentages of participants between treatment groups and their 95% confidence intervals (CIs) were calculated based on an unconditional exact method using 2 inverted 1-sided tests

4. Secondary Outcome: Percentage of Participants Experiencing Grades 1 Through 4 Adverse Events After Switch to E/C/F/TAF or F/R/TAF Throughout the Study and During Coadministeration With LDV/SOF Treatment
Time Frame: Up to 32 weeks plus 30 days
Population: Safety Analysis Set (Whole Study): participants who were randomized into the study and received at least 1 dose of study drug (E/C/F/TAF, F/R/TAF, or LDV/SOF).
  Safety Analysis Set (Part 2): participants who entered Part 2 of the study and received at least one dose of study drug LDV/SOF.
Measure: Number; unit: percentage of participants
Groups:
- E/C/F/TAF + LDV/SOF (Co-administration: Week 8 to Week 20): In Part 2 of the study, participants from part 1 continued receiving E/C/F/TAF 150/150/200/10 mg orally once daily with food until the end of the study and received LDV/SOF 90/400 mg orally once daily with or without food for 12 weeks (until Week 20).
- F/R/TAF + LDV/SOF (Co-administration: Week 8 to Week 20): In Part 2 of the study, participants from part 1 continued receiving (F/R/TAF) 200/25/25 mg orally once daily with food until the end of the study and received LDV/SOF 90/400 mg orally once daily with or without food for 12 weeks (until Week 20).
- E/C/F/TAF + LDV/SOF (Whole Study: Day 1 to Post-HCV Week 12): Part 1: Participants received E/C/F/TAF 150/150/200/10 mg tablet orally once daily with food for 8 weeks.
  Part 2: Participants continued receiving E/C/F/TAF 150/150/200/10 mg tablet orally once daily with food until the end of the study and received LDV/SOF 90/400 mg orally once daily with or without food for 12 weeks (until Week 20).
- F/R/TAF + LDV/SOF (Whole Study: Day 1 to Post-HCV to Week 12): Part 1: Participants received F/R/TAF 200/25/25 mg tablet orally once daily with food for 8 weeks.
  Part 2: Participants continued receiving (F/R/TAF) 200/25/25 mg tablet orally once daily with food until the end of the study and received LDV/SOF 90/400 mg orally once daily with or without food for 12 weeks (until Week 20).
Arm/Group | E/C/F/TAF + LDV/SOF (Co-administration: Week 8 to Week 20) | F/R/TAF + LDV/SOF (Co-administration: Week 8 to Week 20) | E/C/F/TAF + LDV/SOF (Whole Study: Day 1 to Post-HCV Week 12) | F/R/TAF + LDV/SOF (Whole Study: Day 1 to Post-HCV to Week 12)
Number analyzed (Participants) | 72 | 72 | 74 | 74
percentage of participants | 62.5 | 69.4 | 83.8 | 79.7

ADVERSE EVENTS:
Time Frame: Up to 32 weeks plus 30 days
Description: Safety Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug (E/C/F/TAF, F/R/TAF, or LDV/SOF).
Arm/Group | E/C/F/TAF + LDV/SOF | F/R/TAF + LDV/SOF
All-Cause Mortality (participants affected / at risk) | 0/74 | 1/74
Serious Adverse Events (participants affected / at risk) | 7/74 | 12/74
Other Adverse Events (participants affected / at risk) | 46/74 | 36/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E/C/F/TAF + LDV/SOF (N=74) | F/R/TAF + LDV/SOF (N=74)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Testicular abscess (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood pressure orthostatic abnormal (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E/C/F/TAF + LDV/SOF (N=74) | F/R/TAF + LDV/SOF (N=74)
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 3
Nausea (Gastrointestinal disorders) | 4 | 6
Fatigue (General disorders) | 4 | 5
Influenza like illness (General disorders) | 4 | 0
Bronchitis (Infections and infestations) | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 9 | 5
Urinary tract infection (Infections and infestations) | 10 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 1
Headache (Nervous system disorders) | 3 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Hypertension (Vascular disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (4):
  • Study Protocol: Original (2015-12-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT02707601/Prot_000.pdf
  • Study Protocol: Amendment 1 (2016-05-27): https://cdn.clinicaltrials.gov/large-docs/01/NCT02707601/Prot_001.pdf
  • Study Protocol: Amendment 2 (2016-11-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT02707601/Prot_002.pdf
  • Statistical Analysis Plan (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT02707601/SAP_003.pdf